CLINICAL TRIAL: NCT00264511
Title: Does Hyperbaric Oxygen Reduce Complications and Improve Outcomes After Open Tibial Fractures With Severe Soft Tissue Injury? An International Multi-centre Randomized Controlled Trial.
Brief Title: Hyperbaric Oxygen in Lower Leg Trauma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Monash University (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 206/04
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Tibial Fracture; Soft Tissue Injury
Keywords: Hyperbaric oxygen; Crush injury; Tibial fracture; Gustillo 3; soft tissue injury; complications; outcomes; randomised controlled trial
MeSH Terms: conditions — Tibial Fractures; Soft Tissue Injuries; Crush Injuries | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Surgeons initially operating were unaware of allocation. Outcomes arbitrations were conducted by surgeons blind to intervention allocation. Chief investigator masked until follow up data finally received and records locked.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperbaric oxygen treatment (Experimental): Subjects in the HBO treatment group will receive a course of hyperbaric oxygen therapy (HBO) in addition to normal trauma and general care. A total of 12 HBO sessions will be delivered over approximately 8 days. HBO treatment will be provided at 2.4 atmospheres absolute (ATA) pressure for approximately 90 minutes of oxygen therapy. Treatments should be twice daily for the first three days. Minor variability will be allowed with respect to timing and profile of each session.
  Interventions: Other: Hyperbaric Oxygen Treatment
- No hyperbaric oxygenation (No Intervention): Patients randomised to this group will receive standard trauma care.

INTERVENTIONS:
Other: Hyperbaric Oxygen Treatment — Subjects in the HBO treatment group will receive a course of hyperbaric oxygen therapy (HBO) in addition to normal trauma and general care. A total of 12 HBO sessions will be delivered over approximately 8 days. HBO treatment will be provided at 2.4 atmospheres absolute (ATA) pressure for approximately 90 minutes of oxygen therapy. Treatments should be twice daily for the first three days. Minor variability will be allowed with respect to timing and profile of each session.
  Other Names: Hyperbaric oxygen therapy; Hyperbaric Oxygen
  Arms: Hyperbaric oxygen treatment

SUMMARY:
Study hypothesis :Hyperbaric Oxygen may prevent complications and improve outcomes in severe lower limb trauma. We propose to investigate this hypothesis by conducting an International multi centre randomised control trial of standard trauma/orthopaedic care with or without a concurrent course of hyperbaric oxygen treatments.

DETAILED DESCRIPTION:
A randomised controlled trial was undertaken on using hyperbaric oxygen in addition to standard orthopaedic trauma care in severe lower leg injury, defined as an open tibial fracture with severe soft tissue injury. The control arm subjects received standard hospital trauma care whilst the intervention group received standard trauma care with the addition of hyperbaric oxygen therapy with the aim of providing 12 HBOT sessions over the first 9 days of hospital care. The primary outcome measure was the incidence of wound necrosis AND/OR wound infection as assessed at Day 14, with secondary outcomes of wound closure, wound complications, infections and delayed bone union at 12 months plus quality of life and functional questionnaire outcomes at 12 months and 2 years.

The detailed study protocol was published in in June 2015 and the results were published in September 2022. Both publications are Open Access (See References section for publication details)

ELIGIBILITY:
Inclusion Criteria:

* Acute fracture of the tibia with significant soft tissue injury of Gustilo Grade 3
* Enrolment within 48 hours of injury with expectation of commencement of HBO therapy within 48 hours of injury
* Valid consent

Exclusion Criteria:

* Significant head injury
* Injuries incompatible with HBO
* resuscitation requirements incompatible with HBO
* follow up not possible
* hyperbaric contra indications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-02-13; Primary Completion 2014-08-18 (Actual); Study Completion 2016-03-23 (Actual)

PRIMARY OUTCOMES:
Acute phase complication rate | up to 14 days post trauma
  The incidence of acute complications after injury. A composite measure defined as the occurrence within two weeks of trauma of one or both of: significant soft tissue necrosis developing after the initial surgery or significant wound infection.

SECONDARY OUTCOMES:
Amputation rate | 3, 6, 9, 12, 18 and 24 months post trauma
  operative procedure records of a limb amputation related to the trauma under study
Late infection | 3, 6, 9, 12, 18 and 24 months post trauma
  records of diagnosis of wound infection or osteomyelitis or implant infection at defined times
Radiological union | 3, 6, 9, 12, 18 and 24 months post trauma
  electronic image copies of radiographs recorded by treating hospitals
Quality of life score | 3, 6, 9, 12, 18 and 24 months post trauma
  Short Form 36 quality of life questionnaire (algorithm produces a score in the range of 0-100 with higher score better)
Functional outcome score | 3, 6, 9, 12, 18 and 24 months post trauma
  lower limb function component of Short Musculoskeletal Function Assessment ((each question is scored 1-5 with lower score better)
Pain score | 3, 6, 9, 12, 18 and 24 months post trauma
  Subjects self reported pain using a 0-10 visual analogue scale
Delayed union of fracture | 12 months post trauma
  Any diagnosis of delayed union or non union or performance or scheduling of bone graft for union problems
Wound persistence | 3, 6, 9, 12, 18 and 24 months post trauma
  A record of whether any injury related wound remains open at review. Excludes new surgical wounds.
Problem Wounds | 12 months post trauma
  Blinded evaluation of whether post traumatic wounds met the criteria for "Problem Wounds" as a result of requiring readmission to hospital, prolonged wound care, additional surgery or antibiotics that complicated or deteriorated patient recovery

CONTACTS AND LOCATIONS:
Overall Officials: Ian L Millar, MBBS, Study Chair — Bayside Health; Owen Williamson, Principal Investigator — Monash University; Peter Cameron, Principal Investigator — Monash University
Locations (10):
- John Muir Clinical Research Center, Concord, California, United States
- Australia (2):
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Alfred, Melbourne, Victoria
- Universitatsklinikum Graz, Graz, Austria
- Hospital del Trabajador, Santiago, Chile
- City Hospital of Ostrava, Ostrava, Czechia
- Indraprastha Apollo Hospital, New Delhi, Sarita Vihar, India
- Policlinico Umberto 1, University of Rome, Rome, Italy
- Hospital Pedro Hispano, Senhora da Hora, Matosinhos, Portugal
- Karolinska Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Bouachour G, Cronier P, Gouello JP, Toulemonde JL, Talha A, Alquier P. Hyperbaric oxygen therapy in the management of crush injuries: a randomized double-blind placebo-controlled clinical trial. J Trauma. 1996 Aug;41(2):333-9. doi: 10.1097/00005373-199608000-00023. PMID 8760546
- [Background] Garcia-Covarrubias L, McSwain NE Jr, Van Meter K, Bell RM. Adjuvant hyperbaric oxygen therapy in the management of crush injury and traumatic ischemia: an evidence-based approach. Am Surg. 2005 Feb;71(2):144-51. PMID 16022014
- [Background] Millar IL, McGinnes RA, Williamson O, Lind F, Jansson KA, Hajek M, Smart D, Fernandes T, Miller R, Myles P, Cameron P. Hyperbaric Oxygen in Lower Limb Trauma (HOLLT); protocol for a randomised controlled trial. BMJ Open. 2015 Jun 11;5(6):e008381. doi: 10.1136/bmjopen-2015-008381. PMID 26068515
- [Background] Millar IL, Lind FG, Jansson KA, Hajek M, Smart DR, Fernandes TD, McGinnes RA, Williamson OD, Miller RK, Martin CA, Gabbe BJ, Myles PS, Cameron PA; HOLLT investigator group. Hyperbaric Oxygen for Lower Limb Trauma (HOLLT): an international multi-centre randomised clinical trial. Diving Hyperb Med. 2022 Sep 30;52(3):164-174. doi: 10.28920/dhm52.3.164-174. PMID 36100927
- See also: HOLLT website — https://www.hollt.org/Application/home.aspx